CLINICAL TRIAL: NCT01959139
Title: S1313, A Phase IB/II Randomized Study of Modified FOLFIRINOX + Pegylated Recombinant Human Hyaluronidase (PEGPH20) Versus Modified FOLFIRINOX Alone in Patients With Good Performance Status Metastatic Pancreatic Adenocarcinoma
Brief Title: S1313, PEGPH20 in Treating Patients With Newly Diagnosed Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1313; NCI-2013-01776 (Other: NCI); U10CA180888 (NIH); S1313 (Other: SWOG)
Record Dates: First submitted 2013-09-30; First posted 2013-10-09 (Estimated); Results first posted 2020-02-12 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
MeSH Terms: interventions — PEGPH20; Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase II: mFOLFIRINOX (Active Comparator): Patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and irinotecan hydrochloride IV over 1.5 hours on day 2, and 5-fluorouracil (5-FU) IV over 46 hours on days 2-4. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Oxaliplatin; Drug: Leucovorin; Drug: Irinotecan; Drug: 5-fluorouracil
- Phase II: mFOLFIRINOX + PEGPH20 (Experimental): Patients receive pegylated recombinant human hyaluronidase (PEGPH20) IV over 10 minutes on day 1 and oxaliplatin, leucovorin calcium, irinotecan hydrochloride, and 5-fluorouracil (5-FU) as in Arm I. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: PEGPH20; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Irinotecan; Drug: 5-fluorouracil
- Phase I (Experimental): PEGPH20, 3 ug/kg on Day 1 and Day 3/4, IV over 15 minutes; Oxaliplatin, 85 mg/m^2, on Day 2, IV over 2 hours; Leucovorin, 400 mg/m^2, on Day 2, IV over 2 hours; Irinotecan, 180 mg/m^2, on Day 2, IV over 1.5 hours; 5-fluorouracil (5-FU), 2,400 mg/m^2, Days 2-4, IV over 46 hours
  Interventions: Drug: PEGPH20; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Irinotecan; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: PEGPH20 — 3 ug/kg on Day 1, IV over 15 minutes
  Other Names: Pegylated Recombinant Human Hyaluronidase
  Arms: Phase I; Phase II: mFOLFIRINOX + PEGPH20
Drug: Oxaliplatin — 85 mg/m^2, on Day 2, IV over 2 hours
  Other Names: Eloxatin; NSC-266046
Drug: Leucovorin — 400 mg/m^2, on Day 2, IV over 2 hours
  Other Names: leucovorin calcium
Drug: Irinotecan — 180 mg/m^2, on Day 2, IV over 1.5 hours
  Other Names: CPT-11; NSC-616348
Drug: 5-fluorouracil — 2,400 mg/m^2, Days 2-4, IV over 46 hours
  Other Names: 5-FU; Adrucil; NSC-19893

SUMMARY:
This partially randomized phase I/II trial studies the side effects and best dose of pegylated recombinant human hyaluronidase (PEGPH20) when given together with combination chemotherapy and to see how well they work compared with combination chemotherapy alone in treating patients with newly diagnosed pancreatic cancer that has spread to other places in the body. Pegylated recombinant human hyaluronidase may help chemotherapy drugs work better by making tumor cells more sensitive to the drugs. Drugs used in chemotherapy, such as leucovorin calcium, fluorouracil, irinotecan hydrochloride, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether combination chemotherapy is more effective with or without pegylated recombinant human hyaluronidase in treating pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of modified leucovorin calcium, fluorouracil, irinotecan hydrochloride and oxaliplatin (mFOLFIRINOX) in combination with PEGPH20 and select the optimal dose of PEGPH20 for the phase II portion in patients with metastatic pancreatic adenocarcinoma. (Phase I) II. To assess the overall survival of patients with metastatic pancreatic adenocarcinoma treated with mFOLFIRINOX + PEGPH20 compared to those treated with mFOLFIRINOX alone. (Phase II)

SECONDARY OBJECTIVES:

I. To assess progression free survival (PFS) in patients receiving mFOLFIRINOX with PEGPH20 and patients receiving mFOLFIRINOX alone in this patient population.

II. To assess objective tumor response (confirmed and unconfirmed, complete and partial) in patients with measurable disease treated with mFOLFIRINOX with PEGPH20 and patients receiving mFOLFIRINOX alone in this patient population.

III. To determine the frequency, severity, and tolerability of adverse events of mFOLFIRINOX with PEGPH20.

TERTIARY OBJECTIVES:

I. To explore the correlation of maximum decrease in cancer antigen (CA) 19-9 levels and time to maximum decrease in CA 19-9 levels with overall survival, progression-free survival and response.

II. To explore the correlation of plasma hyaluronan (HA) and tumor expression of HA with overall survival, progression-free survival and response.

OUTLINE: This is a phase I, dose de-escalation study of pegylated recombinant human hyaluronidase followed by a randomized phase II study.

PHASE I: Patients receive pegylated recombinant human hyaluronidase intravenously (IV) over 10 minutes on day 1*; oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and irinotecan hydrochloride IV over 1.5 hours on day 2; and fluorouracil IV over 46 hours on days 2-4. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and irinotecan hydrochloride IV over 1.5 hours on day 2, and fluorouracil IV over 46 hours on days 2-4. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive pegylated recombinant human hyaluronidase IV over 10 minutes on day 1* and oxaliplatin, leucovorin calcium, irinotecan hydrochloride, and fluorouracil as in Arm I. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

*NOTE: Some patients also receive pegylated recombinant human hyaluronidase on day 3 or 4 of courses 1 and 2.

After completion of study treatment, patients are followed up for 3 years.

ELIGIBILITY:
* Patients must have newly diagnosed, untreated metastatic histologically or cytologically documented pancreatic adenocarcinoma; patients must not have known history of brain metastases
* Patients must have measurable metastatic disease; computed tomography (CT) scans or magnetic resonance imaging (MRI)s used to assess measurable disease must have been completed within 28 days prior to registration; CT scans or MRIs used to assess non-measurable disease must have been completed within 42 days prior to registration; CT scans or MRIs must be assessed and documented on the Baseline Tumor Assessment Form (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1)
* Patients must not have had any prior treatment with oxaliplatin or irinotecan within 3 years prior to registration; patients must not have had prior chemotherapy in metastatic setting; prior abdominal radiation therapy is not allowed
* Patients must have a Zubrod performance status of 0-1
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) both =< 2.5 X IULN in the absence of liver metastases or =< 5.0 x IULN with liver metastasis
* Serum albumin >= 3 g/dL
* Serum creatinine =< ULN within 14 days prior to registration OR calculated creatinine clearance > 50 ml/min; the serum creatinine value used in the calculation must have been obtained within 14 days prior to registration
* Patients must have international normalized ratio (INR) =< 1.2 within 14 days prior to registration; patients must not be receiving warfarin for therapeutic use, have history of cerebrovascular accident (CVA), history of transient ischemic attack (TIA) requiring intervention or treatment, pre-existing carotid artery disease requiring intervention or treatment, or current use of megestrol acetate (use within 10 days of registration)
* Patients must not be receiving chronic treatment (equivalent of prednisone > 10 mg/day) with systemic steroids or other immuno-suppressive agent
* Patients must not have liver disease such a cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* Patients must not have active bleeding or a pathological condition that is associated with a high risk of bleeding
* Patients with a known history of human immunodeficiency virus (HIV) must not be on active treatment for HIV
* Patients must have no non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with protocol therapy
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Patients must have tumor (paraffin block or slides) available for submission and be willing to submit tumor and blood samples
* Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* Patients planning to enroll in the phase I portion of this study must first have a slot reserved in advance of the registration; all site staff will use OPEN to create a slot reservation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-01-23 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh K Ramanathan, M.D., Study Chair — Virginia G. Piper Cancer Center
Locations (154):
- United States (154):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - City of Hope Corona, Corona, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - City of Hope West Covina, West Covina, California
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Medical Oncology and Hematology Group PC-Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Charlotte Hungerford Hospital Center for Cancer Care, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Randolph Hospital, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington

REFERENCES:
- [Derived] Ramanathan RK, McDonough SL, Philip PA, Hingorani SR, Lacy J, Kortmansky JS, Thumar J, Chiorean EG, Shields AF, Behl D, Mehan PT, Gaur R, Seery T, Guthrie KA, Hochster HS. Phase IB/II Randomized Study of FOLFIRINOX Plus Pegylated Recombinant Human Hyaluronidase Versus FOLFIRINOX Alone in Patients With Metastatic Pancreatic Adenocarcinoma: SWOG S1313. J Clin Oncol. 2019 May 1;37(13):1062-1069. doi: 10.1200/JCO.18.01295. Epub 2019 Feb 28. PMID 30817250

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 126 participants were enrolled to this study, however, 1 withdrew consent and 3 were ineligible.
Groups:
- Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 and Day 3/4: PEGPH20, 3 ug/kg on Day 1 and Day 3/4, IV over 15 minutes;
  Oxaliplatin, 85 mg/m^2, on Day 2, IV over 2 hours;
  Leucovorin, 400 mg/m^2, on Day 2, IV over 2 hours;
  Irinotecan, 180 mg/m^2, on Day 2, IV over 1.5 hours;
  5-fluorouracil (5-FU), 2,400 mg/m^2, Days 2-4, IV over 46 hours
- Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 Only: PEGPH20: 3 ug/kg on Day 1, IV over 15 minutes
  Oxaliplatin: 85 mg/m^2, on Day 2, IV over 2 hours
  Leucovorin: 400 mg/m^2, on Day 2, IV over 2 hours
  Irinotecan: 180 mg/m^2, on Day 2, IV over 1.5 hours
  5-fluorouracil: 2,400 mg/m^2, Days 2-4, IV over 46 hours
Period: Phase I: Cohort 1
Arm/Group | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 and Day 3/4 | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 Only | Phase II: mFOLFIRINOX | Phase II: mFOLFIRINOX + PEGPH20
Started | 5 | 0 | 0 | 0
Completed | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase I: Cohort 2
Arm/Group | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 and Day 3/4 | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 Only | Phase II: mFOLFIRINOX | Phase II: mFOLFIRINOX + PEGPH20
Started | 0 | 6 | 0 | 0
Completed | 0 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase II
Arm/Group | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 and Day 3/4 | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 Only | Phase II: mFOLFIRINOX | Phase II: mFOLFIRINOX + PEGPH20
Started | 0 | 0 | 56 | 55
Assessed for AEs | 0 | 0 | 54 | 51
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 56 | 55
Not completed — Disease progression | 0 | 0 | 26 | 34
Not completed — Adverse Event | 0 | 0 | 10 | 11
Not completed — Patient Refusal | 0 | 0 | 5 | 4
Not completed — Death | 0 | 0 | 3 | 1
Not completed — Other/Unknown | 0 | 0 | 8 | 5
Not completed — On treatment | 0 | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 and Day 3/4 | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 Only | Phase II: mFOLFIRINOX | Phase II: mFOLFIRINOX + PEGPH20 | Total
Number analyzed (Participants) | 5 | 6 | 56 | 55 | 122
Age, Continuous [Median (Full Range); unit: years] | 65.4 [41.1 to 72.4] | 60.2 [49.7 to 72.9] | 60.5 [31.9 to 74.9] | 63.9 [40.4 to 73.8] | 62.2 [31.9 to 74.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 25 | 31 | 61
  Male | 2 | 4 | 31 | 24 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 4 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 4 | 1 | 7
  White | 3 | 4 | 46 | 43 | 96
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 4 | 7
Zubrod performance status [Count of Participants; unit: Participants] — Scale: 0-5, with 0 denoting perfect health and 5 death.
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1: Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    0 | 2 | 5 | 31 | 32 | 70
    1 | 3 | 1 | 25 | 23 | 52
Primary site [Count of Participants; unit: Participants]
  Head of pancreas | 2 | 4 | 16 | 19 | 41
  Body of pancreas | 1 | 0 | 16 | 16 | 33
  Tail of pancreas | 2 | 1 | 15 | 11 | 29
  Pancreas, NOS | 0 | 1 | 9 | 9 | 19
Sites of involvement [Count of Participants; unit: Participants]
  Primary tumor/pancreas | 4 | 4 | 51 | 49 | 108
  Regional lymph nodes | 3 | 3 | 22 | 16 | 44
  Distant lymph nodes | 0 | 3 | 6 | 5 | 14
  Lung | 1 | 1 | 18 | 14 | 34
  Liver | 4 | 3 | 45 | 42 | 94
  Peritoneum | 1 | 1 | 12 | 11 | 25
  Other | 1 | 1 | 12 | 9 | 23
Serum cancer antigen (CA) 19-9 [Count of Participants; unit: Participants]
  < 37 | 1 | 1 | 10 | 7 | 19
  >= 37 | 4 | 5 | 46 | 48 | 103
Prior treatment for pancreatic cancer [Count of Participants; unit: Participants]
  Chemotherapy | 0 | 1 | 3 | 4 | 8
  Surgery | 0 | 1 | 2 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of PEGPH20 in Combination With mFOLFIRINOX
Description: Assess safety of mFOLFIRINOX in combination with PEGPH20 and select the optimal dose of PEGPH20 for the Phase II portion.
  MTD of PEGPH20 in combination with mFOLFORINOX was evaluated by testing decreasing doses of PEGPH20 from 3mcg/kg on Day 1 and Day 3/4, to 3mcg/kg on Day 1 only and to 1.6 mcg/kg on Day 1 only.
  MTD reflects the highest dose that had a dose-limiting toxicity (DLT) rate of ≤ 17%. DLTs were defined as treatment regimen related: grade ≥ 3 non-hematologic toxicity; grade 4 absolute neutrophil count (ANC) anemia or thrombocytopenia; grade 4 ANC lasting > 7 days; grade ≥ 3 febrile neutropenia; grade ≥ 3 elevation of aspartate aminotransferase (AST)/alanine aminotransferase (ALT), total bilirubin, and creatinine; delay in starting the 2nd cycle of mFOLFIRINOX by > 2 weeks due to drug related toxicity.
  DLT were graded using the NCI CTCAE version 4. Note: the third and lowest dose level was not reached.
Time Frame: 2 cycles of 14 days
Population: All analyzable patients who experienced a dose limiting toxicity attributable to PEGPH20 and/or mFOLFIRINOX in the first cycle
Measure: Number; unit: ug/kg
Groups:
- Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1: PEGPH20: 3 ug/kg on Day 1, IV over 15 minutes
  Oxaliplatin: 85 mg/m^2, on Day 2, IV over 2 hours
  Leucovorin: 400 mg/m^2, on Day 2, IV over 2 hours
  Irinotecan: 180 mg/m^2, on Day 2, IV over 1.5 hours
  5-fluorouracil: 2,400 mg/m^2, Days 2-4, IV over 46 hours
- All Phase 1 Participants: Phase I participants that received PEGPH20 at the assigned dose for cycle 1.
Arm/Group | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 and Day 3/4 | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 | All Phase 1 Participants
Number analyzed (Participants) | 5 | 6 | 11
ug/kg | 0 | 3 | 3

2. Primary Outcome: Phase II: Overall Survival
Description: Time from date of registration to date of death due to any cause. Participants last known to be alive are censored at date of last contact.
  Assessed using the logrank test.
Time Frame: From date of registration to date of death due to any cause, assessed up to 3 years
Population: Eligible and analyzable participants
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase II: mFOLFIRINOX: Participants receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and irinotecan hydrochloride IV over 1.5 hours on day 2, and 5-fluorouracil (5-FU) IV over 46 hours on days 2-4. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Oxaliplatin: 85 mg/m^2, on Day 2, IV over 2 hours
  Leucovorin: 400 mg/m^2, on Day 2, IV over 2 hours
  Irinotecan: 180 mg/m^2, on Day 2, IV over 1.5 hours
  5-fluorouracil: 2,400 mg/m^2, Days 2-4, IV over 46 hours
- Phase II: mFOLFIRINOX + PEGPH20: Participants receive pegylated recombinant human hyaluronidase (PEGPH20) IV over 10 minutes on day 1 and oxaliplatin, leucovorin calcium, irinotecan hydrochloride, and 5-fluorouracil (5-FU) as in Arm I. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  PEGPH20: 3 ug/kg on Day 1, IV over 15 minutes
  Oxaliplatin: 85 mg/m^2, on Day 2, IV over 2 hours
  Leucovorin: 400 mg/m^2, on Day 2, IV over 2 hours
  Irinotecan: 180 mg/m^2, on Day 2, IV over 1.5 hours
  5-fluorouracil: 2,400 mg/m^2, Days 2-4, IV over 46 hours
Arm/Group | Phase II: mFOLFIRINOX | Phase II: mFOLFIRINOX + PEGPH20
Number analyzed (Participants) | 56 | 55
months | 14.4 [9.2 to 18.0] | 7.7 [4.5 to 10.7]
Statistical Analysis 1: Comparison: Phase II: mFOLFIRINOX vs Phase II: mFOLFIRINOX + PEGPH20; Test type: Superiority; p < 0.01, Regression, Cox; Hazard Ratio (HR) = 2.07, 95% CI 2-sided [1.28 to 3.34]

3. Secondary Outcome: Progression Free Survival (PFS) (Phase II)
Description: Time from date of registration to date of first documentation of progression or symptomatic deterioration or death due to any cause. Participants last known to be alive without report of progression are censored at date of last contact.
Time Frame: From date of registration to date of death due to any cause, assessed up to 3 years
Population: Eligible and analyzable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: mFOLFIRINOX | Phase II: mFOLFIRINOX + PEGPH20
Number analyzed (Participants) | 56 | 55
months | 6.2 [3.7 to 10.2] | 4.3 [2.4 to 5.8]
Statistical Analysis 1: Comparison: Phase II: mFOLFIRINOX vs Phase II: mFOLFIRINOX + PEGPH20; Test type: Superiority; p = 0.01, Regression, Cox; Hazard Ratio (HR) = 1.74, 95% CI 2-sided [1.14 to 2.66]

4. Secondary Outcome: Objective Tumor Response Rate (Confirmed and Unconfirmed, Complete and Partial)
Description: Objective tumor response rate (complete response, unconfirmed complete response, partial response, unconfirmed partial response) in patients with measurable disease were assessed in each arm and compared between arms using Chi-squared test.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions
Time Frame: Up to 3 years
Population: Participants with measurable disease
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Phase II: mFOLFIRINOX | Phase II: mFOLFIRINOX + PEGPH20
Number analyzed (Participants) | 56 | 55
percent of participants | 45 [32 to 58] | 33 [20 to 45]

5. Secondary Outcome: Number of Patients With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 4.0. Only adverse events that are possibly, probably or definitely related to study drug are reported.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living e.g. bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.
  Grade 4: Life-threatening consequences; urgent intervention indicated.
  Grade 5: Death related to adverse event
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Population: Patients who received at least one dose of protocol treatment. Only 105 participants in the phase II trial were assessed for AEs, as 6 participants did not receive protocol treatment.
Measure: Number; unit: Participants
Groups:
- Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 and Day 3/4: PEGPH20, 3 ug/kg on Day 1 and Day 3/4, IV over 15 minutes__Oxaliplatin, 85 mg/m^2, on Day 2, IV over 2 hours__Leucovorin, 400 mg/m^2, on Day 2, IV over 2 hours__Irinotecan, 180 mg/m^2, on Day 2, IV over 1.5 hours__5-fluorouracil (5-FU), 2,400 mg/m^2, Days 2-4, IV over 46 hours
- Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 Only: PEGPH20: 3 ug/kg on Day 1, IV over 15 minutes__Oxaliplatin: 85 mg/m^2, on Day 2, IV over 2 hours__Leucovorin: 400 mg/m^2, on Day 2, IV over 2 hours__Irinotecan: 180 mg/m^2, on Day 2, IV over 1.5 hours__5-fluorouracil: 2,400 mg/m^2, Days 2-4, IV over 46 hours
- Phase II: mFOLFIRINOX: Participants receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and irinotecan hydrochloride IV over 1.5 hours on day 2, and 5-fluorouracil (5-FU) IV over 46 hours on days 2-4. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.__Oxaliplatin: 85 mg/m^2, on Day 2, IV over 2 hours__Leucovorin: 400 mg/m^2, on Day 2, IV over 2 hours__Irinotecan: 180 mg/m^2, on Day 2, IV over 1.5 hours__5-fluorouracil: 2,400 mg/m^2, Days 2-4, IV over 46 hours
- Phase II: PEGPH20 + mFOLFIRINOX: Participants receive pegylated recombinant human hyaluronidase (PEGPH20) IV over 10 minutes on day 1 and oxaliplatin, leucovorin calcium, irinotecan hydrochloride, and 5-fluorouracil (5-FU) as in Arm I. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.__PEGPH20: 3 ug/kg on Day 1, IV over 15 minutes__Oxaliplatin: 85 mg/m^2, on Day 2, IV over 2 hours__Leucovorin: 400 mg/m^2, on Day 2, IV over 2 hours__Irinotecan: 180 mg/m^2, on Day 2, IV over 1.5 hours__5-fluorouracil: 2,400 mg/m^2, Days 2-4, IV over 46 hours
Arm/Group | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 and Day 3/4 | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 Only | Phase II: mFOLFIRINOX | Phase II: PEGPH20 + mFOLFIRINOX
Number analyzed (Participants) | 5 | 6 | 54 | 51
Participants
  Abdominal pain | 0 | 0 | 1 | 3
  Acute kidney injury | 1 | 0 | 0 | 0
  Alanine aminotransferase increased | 1 | 1 | 0 | 3
  Alkaline phosphatase increased | 0 | 1 | 0 | 2
  Anemia | 0 | 0 | 4 | 2
  Anorexia | 0 | 0 | 2 | 3
  Arthralgia | 0 | 0 | 0 | 1
  Ascites | 0 | 0 | 0 | 1
  Aspartate aminotransferase increased | 0 | 1 | 0 | 0
  Blood bilirubin increased | 1 | 0 | 0 | 1
  Creatinine increased | 0 | 0 | 1 | 0
  Dehydration | 1 | 1 | 7 | 4
  Depression | 0 | 0 | 1 | 0
  Diarrhea | 1 | 0 | 10 | 12
  Esophagitis | 0 | 0 | 0 | 1
  Fatigue | 2 | 1 | 6 | 11
  Febrile neutropenia | 0 | 0 | 1 | 0
  Gallbladder obstruction | 1 | 0 | 0 | 0
  Gastrointestinal disorders - Other, specify | 0 | 0 | 0 | 1
  General disorders and admin site conditions- Other | 0 | 0 | 1 | 0
  Generalized muscle weakness | 0 | 0 | 1 | 3
  Hyperglycemia | 0 | 0 | 1 | 1
  Hypertension | 0 | 0 | 1 | 0
  Hypokalemia | 1 | 1 | 3 | 4
  Hyponatremia | 1 | 1 | 1 | 3
  Hypophosphatemia | 0 | 0 | 0 | 1
  Hypotension | 0 | 1 | 0 | 0
  Infections and infestations - Other, specify | 0 | 0 | 1 | 0
  Infusion related reaction | 0 | 0 | 0 | 1
  Leukocytosis | 0 | 0 | 2 | 1
  Lung infection | 0 | 0 | 1 | 0
  Lymphocyte count decreased | 0 | 0 | 1 | 4
  Mucositis oral | 1 | 0 | 0 | 4
  Myalgia | 1 | 0 | 0 | 2
  Nausea | 1 | 0 | 8 | 12
  Neutrophil count decreased | 0 | 0 | 4 | 3
  Pain | 0 | 0 | 1 | 0
  Paresthesia | 0 | 0 | 1 | 0
  Peripheral motor neuropathy | 0 | 0 | 1 | 1
  Peripheral sensory neuropathy | 0 | 2 | 2 | 5
  Peritoneal infection | 0 | 0 | 0 | 1
  Platelet count decreased | 0 | 1 | 2 | 3
  Portal vein thrombosis | 0 | 0 | 0 | 1
  Pulmonary hypertension | 0 | 0 | 1 | 0
  Resp, thoracic and mediastinal disorders - Other | 0 | 0 | 1 | 0
  Sepsis | 1 | 0 | 1 | 1
  Skin infection | 0 | 0 | 0 | 1
  Small intestine infection | 0 | 0 | 0 | 1
  Spasticity | 0 | 0 | 0 | 1
  Thromboembolic event | 0 | 0 | 1 | 5
  Ventricular tachycardia | 0 | 0 | 1 | 0
  Vomiting | 1 | 1 | 8 | 10
  Weight loss | 0 | 0 | 1 | 0
  White blood cell decreased | 0 | 0 | 2 | 2

6. Other Pre Specified Outcome: Cancer Antigen (CA) 19-9 Levels
Description: Explore correlation of maximum decrease in CA 19-9 levels to maximum decrease in CA 19-9 levels with overall survival, progression-free survival and response.
Time Frame: Within 2 years of the end of the study
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Plasma Expression of Hyaluronan (HA)
Time Frame: Within 2 years of end of study
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Tumor Expression of HA
Time Frame: Within 2 years of end of study
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Description: Only 105 participants in the phase II trial were assessed for AEs, as 6 participants did not receive protocol therapy.
Arm/Group | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 and Day 3/4 | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 Only | Phase II: mFOLFIRINOX | Phase II: PEGPH20 + mFOLFIRINOX
All-Cause Mortality (participants affected / at risk) | 5/5 | 5/6 | 49/56 | 50/55
Serious Adverse Events (participants affected / at risk) | 3/5 | 4/6 | 9/54 | 36/51
Other Adverse Events (participants affected / at risk) | 4/5 | 6/6 | 52/54 | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 and Day 3/4 (N=5) | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 Only (N=6) | Phase II: mFOLFIRINOX (N=54) | Phase II: PEGPH20 + mFOLFIRINOX (N=51)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 6
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 1 | 7
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 9
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 2 | 9
Death NOS (General disorders) | 0 | 0 | 1 | 1
Fatigue (General disorders) | 1 | 1 | 0 | 5
Fever (General disorders) | 0 | 0 | 0 | 1
Infusion related reaction (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0 | 1
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatobiliary disorders-Other (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Peritoneal infection (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1 | 2
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Small intestine infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Weight loss (Investigations) | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 3
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2
Transient ischemic attacks (Nervous system disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 1 | 4 | 11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 and Day 3/4 (N=5) | Phase I: mFOLFIRINOX + PEGPH20, 3 ug/kg on Day 1 Only (N=6) | Phase II: mFOLFIRINOX (N=54) | Phase II: PEGPH20 + mFOLFIRINOX (N=51)
Anemia (Blood and lymphatic system disorders) | 1 | 4 | 36 | 37
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 3 | 2
Cardiac disorders-Other (Cardiac disorders) | 0 | 0 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1 | 3
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 3
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2 | 0
Endocrine disorders-Other (Endocrine disorders) | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Blurred vision (Eye disorders) | 2 | 1 | 6 | 2
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Eye disorders-Other (Eye disorders) | 0 | 0 | 1 | 3
Eye pain (Eye disorders) | 1 | 0 | 0 | 2
Floaters (Eye disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 27 | 22
Anal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Anal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Bloating (Gastrointestinal disorders) | 1 | 1 | 4 | 6
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 4 | 20 | 16
Diarrhea (Gastrointestinal disorders) | 4 | 4 | 41 | 38
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 2 | 5
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 8 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 3 | 4
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Esophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 8 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 1 | 0 | 4 | 4
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastroparesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 1 | 10 | 11
Nausea (Gastrointestinal disorders) | 2 | 4 | 39 | 39
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral dysesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 26 | 23
Chills (General disorders) | 0 | 0 | 6 | 1
Edema face (General disorders) | 0 | 0 | 1 | 0
Edema limbs (General disorders) | 2 | 2 | 10 | 20
Edema trunk (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 4 | 5 | 42 | 40
Fever (General disorders) | 0 | 1 | 7 | 2
Flu like symptoms (General disorders) | 1 | 0 | 1 | 1
Gait disturbance (General disorders) | 0 | 0 | 2 | 0
General disorders and admin site conditions - Other (General disorders) | 0 | 0 | 4 | 4
Infusion related reaction (General disorders) | 1 | 0 | 7 | 8
Localized edema (General disorders) | 0 | 0 | 1 | 1
Malaise (General disorders) | 0 | 0 | 3 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 3
Pain (General disorders) | 1 | 2 | 12 | 10
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Bladder infection (Infections and infestations) | 0 | 0 | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0
Hepatic infection (Infections and infestations) | 0 | 0 | 1 | 0
Infections and infestations-Other (Infections and infestations) | 0 | 0 | 6 | 3
Mucosal infection (Infections and infestations) | 0 | 0 | 3 | 2
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1
Pelvic infection (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 0
Upper respiratory infection (Infections and infestations) | 0 | 2 | 2 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 5 | 4
Vaginal infection (Infections and infestations) | 0 | 0 | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 5
Alanine aminotransferase increased (Investigations) | 2 | 3 | 18 | 19
Alkaline phosphatase increased (Investigations) | 2 | 3 | 24 | 24
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 17 | 18
Blood bilirubin increased (Investigations) | 1 | 0 | 3 | 3
Creatinine increased (Investigations) | 1 | 0 | 1 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1 | 0 | 0
GGT increased (Investigations) | 0 | 0 | 0 | 1
INR increased (Investigations) | 0 | 1 | 1 | 2
Investigations-Other (Investigations) | 0 | 1 | 1 | 4
Lymphocyte count decreased (Investigations) | 1 | 0 | 8 | 7
Lymphocyte count increased (Investigations) | 1 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 2 | 9 | 6
Platelet count decreased (Investigations) | 2 | 2 | 27 | 22
Weight loss (Investigations) | 0 | 3 | 18 | 27
White blood cell decreased (Investigations) | 1 | 2 | 10 | 9
Anorexia (Metabolism and nutrition disorders) | 3 | 3 | 25 | 26
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 15 | 6
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2 | 22 | 24
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 3 | 24 | 26
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 5 | 24
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 5 | 28 | 19
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 6 | 4
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 17 | 18
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 6 | 7
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 13 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 11 | 6
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 6 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 4
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 2 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 1
Concentration impairment (Nervous system disorders) | 0 | 0 | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 9 | 9
Dysarthria (Nervous system disorders) | 1 | 0 | 3 | 2
Dysesthesia (Nervous system disorders) | 1 | 0 | 1 | 2
Dysgeusia (Nervous system disorders) | 3 | 3 | 12 | 13
Facial muscle weakness (Nervous system disorders) | 0 | 0 | 1 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 9 | 5
Memory impairment (Nervous system disorders) | 0 | 1 | 1 | 1
Nervous system disorders-Other (Nervous system disorders) | 0 | 0 | 2 | 2
Paresthesia (Nervous system disorders) | 2 | 0 | 10 | 7
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1 | 2 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 4 | 32 | 24
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Sinus pain (Nervous system disorders) | 0 | 0 | 0 | 1
Spasticity (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 3 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 10 | 5
Confusion (Psychiatric disorders) | 0 | 0 | 2 | 1
Depression (Psychiatric disorders) | 0 | 0 | 7 | 4
Insomnia (Psychiatric disorders) | 1 | 2 | 9 | 10
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 1
Psychiatric disorders-Other (Psychiatric disorders) | 0 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 2 | 2
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 2
Renal calculi (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 6 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 5 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 4
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 4
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 12 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 7 | 5
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 1
Hematoma (Vascular disorders) | 0 | 0 | 1 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 3 | 5
Hypertension (Vascular disorders) | 1 | 0 | 9 | 8
Hypotension (Vascular disorders) | 0 | 1 | 5 | 2
Thromboembolic event (Vascular disorders) | 0 | 0 | 3 | 1
Vascular disorders-Other (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT01959139/Prot_SAP_ICF_000.pdf